CLINICAL TRIAL: NCT01831011
Title: Efficacy and Safety of Mildronate for Acute Ischemic Stroke: a Randomized, Double-blind, Active-controlled Phase II Multicenter Trial
Brief Title: Mildronate for Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: xijing-008
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Acute Ischemic Stroke
Keywords: randomized trial; acute ischemic stroke; mildronate
MeSH Terms: conditions — Ischemic Stroke | interventions — 3-(2,2,2-trimethylhydrazine)propionate; cinepazide; WW Domain-Containing Oxidoreductase; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mildronate (Experimental): infusion of mildronate
  Interventions: Drug: mildronate injection; Drug: aspirin
- cinepazide maleate (Active Comparator): infusion of cinepazide maleate
  Interventions: Drug: cinepazide maleate injection; Drug: aspirin

INTERVENTIONS:
Drug: mildronate injection
  Other Names: infusion of mildronate infusion of mildronate(500mg) once a day and for 14 da
  Arms: mildronate
Drug: cinepazide maleate injection
  Other Names: infusion of plabcebo once a day and for 14 days
  Arms: cinepazide maleate
Drug: aspirin
  Other Names: infusion of aspirin (100mg) once a day for days

SUMMARY:
Mildronate an inhibitor of carnitine-dependent metabolism, is considered an anti-ischemic drug. This study aims to evaluate the efficacy and safety of mildronate injection in treating acute ischemic stroke.

DETAILED DESCRIPTION:
A randomized, double-blind, multi-center clinical study was made on mildronate injection for treating acute cerebral infarction. 113 cases in the experimental group were given with mildronate injection, while 114 cases in the active-control group were given with cinepazide maleate injection. In addition, both groups were given aspirin as basic treatments. Modified Rankin Scale (mRS) score at 2 weeks and 3 months, National Institutes of Health Stroke Scale (NIHSS) score and Barthel Index score at 2 weeks after treatment, vital signs and adverse events were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* (i) had a clinical diagnosis of acute ischaemic stroke ,on the first episode within the previous 7 days, and confirmed on CT or MRI brain imaging.(ii) were between 18 to 80 years of age (patients >= 70 years were not combined with any other poor physical condition except ischaemic stroke )(iii)had a score of 5-22 on the National Institutes of Health Stroke Scale (NIHSS).(iv)had a report that liver and kedney function were less than 1.5 folds of normal value.

Exclusion Criteria:

* (i) had other intracranial pathologies (e.g. cerebral hemorrhage, tumour, infection), (ii) were pregnant or nursing ;(iii) had a neurological or psychiatric disease ;(iv) had significant drug or alcohol misuse, (v)had been given thrombolytic therapy or medication forbidden by study protocol; (vi)participated in a clinical trial in the past 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
the modified Rankin scale | 3 months

SECONDARY OUTCOMES:
NIHSS scores | 15 days
the Barthel index | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, MD, Study Director — the Department of Neurology , Xijing Hospital; Guang Yun Zhang, MD, Principal Investigator — the Department of Neurology , Xijing Hospital; Yi Zhu, MD, Principal Investigator — the Department of Neurology , Xijing Hospital
Locations (1):
- the Department of Neurology, Xi’an, Shanxi, China